CLINICAL TRIAL: NCT06133257
Title: Effects of Goal-Directed Fluid Therapy Guided by Inferior Vena Cava Collapsibility Index on Hemodynamics and Enhanced Recovery in Patients Undergoing Lower Limb Surgeries
Brief Title: Goal-Directed Fluid Therapy in Patients Undergoing Lower Limb Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mahmoud Aboubakr Abdelkader, resident doctor of anesthesia, Intensive Care and Pain Management, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11122
Record Dates: First submitted 2023-10-31; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia; ERAS; Fluid Overload; Hypovolemia; Surgical Shock
MeSH Terms: conditions — Edema; Hypovolemia; Shock, Surgical

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GD Group (Active Comparator): Patients will take oral clear fluids with carbohydrates content 2 hours preoperatively and intraoperative fluid intake will be guided by Inferior vena cava(IVC) diameter.
  Interventions: Procedure: Goal-Directed Fluid Therapy guided by Inferior Vena Cava Collapsibility Index
- C Group (Active Comparator): the standard fluid management group patients will be fasting 6 hours preoperatively and will receive intraoperative fluid in standard manner.
  Interventions: Procedure: standard fluid management

INTERVENTIONS:
Procedure: Goal-Directed Fluid Therapy guided by Inferior Vena Cava Collapsibility Index — Measuring Inferior vena cava(IVC) diameter using ultrasound then calculation Inferior vena cava(IVC) collapsibility index and administer fluid accordingly.
  Arms: GD Group
Procedure: standard fluid management — standard fluid management
  Arms: C Group

SUMMARY:
Controlling the amount of fluids given to patients in perioperative setting can significantly influence their outcomes.

DETAILED DESCRIPTION:
To overcome these problems and avoid the complications of over or underhydration, we use the Goal-directed fluid therapy(GDFT) guided by Inferior vena cava(IVC) collapsibility index approach in which dynamic parameters of volume responsiveness as a guide for fluid therapy. This will ensure that the fluids given were deficient from the circulation and improve the recovery of the patients according to enhanced recovery after surgery(ERAS) protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patient's acceptance.
* Patients planned for elective lower limb surgery under spinal anesthesia.
* Both sexes
* Body Mass Index(BMI): <35
* Age: 21 ~ 65 years
* American Society of Anesthesiologists(ASA) Physical Status Classification System: Class I & II
* Duration of surgery 2~3 hours

Exclusion Criteria:

* Advanced kidney, liver, respiratory or cardiovascular disease.
* Contraindication for spinal anesthesia.
* Patients shifted to general anesthesia for any reason.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Blood Pressure | intraoperatively every 5 minutes
  intraoperative mean arterial blood pressure measured in mmHg
Quality of Recovery-40 score(QoR-40) | 24 hours postoperative
  QoR-40 score ranges from 40 to 200, the higher the score the better the outcome
Heart Rate | intraoperatively every 5 minutes
  intraoperative heart rate will be continuously monitored and recorded every 5 minutes
Post Anesthesia Care Unit(PACU) Stay | 2 hours postoperatively
  time spent in PACU after surgery measured in minutes

SECONDARY OUTCOMES:
Total fluid intake during operation | intraoperatively
  Total fluid intake during operation
Number of patients that needed Ephedrine or Atropine | intraoperatively
  Number of patients that needed Ephedrine or Atropine intraoperatively
Peripheral perfusion index | Intraoperatively
  Peripheral Perfusion Index (PPI) is defined as "the ratio of pulsatile blood flow to the non-pulsatile blood flow". It ranges from 0.02% to 20% and it is measured using specific types pulse oximetry and it reflects the perfusion status of the body.
Length of hospital stay | the patient will be followed up for 60 days from day of surgery
  the number of days from day of surgery until patient's discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdelkader, MBBCh, Principal Investigator — Anesthesia, Intensive Care and Pain Management department, Faculty of Medicine, Zagazig University

IPD SHARING:
Plan to Share IPD: No